CLINICAL TRIAL: NCT07116005
Title: The Influence of Mandala Art Therapy on Practical Examination Anxiety Among Undergraduate Nursing Students
Brief Title: Mandala Art Therapy on Practical Examination Anxiety
Acronym: Mandala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Pouran Varvani Farahani, PhD in Pediatric Nursing, Near East University , Faculty of Nursing, Nicosia, TRNC, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVF2025CAM003
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Exam Anxiety
Keywords: Art Therapy; Exam Anxiety; Complementary Therapies

STUDY DESIGN:
Intervention Model Description: Participants in this clinical trial were randomly assigned to one of two groups:
  an experimental group that participated in Mandala Art Therapy (coloring a Mandala design for 20 minutes prior to the OSCE), and a control group that received standard academic preparation without any additional intervention. Both groups were observed in parallel throughout the study period to assess changes in exam anxiety levels.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-Blind (Investigator, Outcomes Assessor):
  To minimize bias, a double-blind approach is employed. The data are collected by the researcher, who remains unaware of group assignments, and the statistician performing the analysis is also blinded to the allocation. The data are analyzed as anonymous variables (x# and x#) to preserve objectivity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Art Therapy (Experimental): Behavioral: Mandala Coloring Participants in this group receive the Mandala Art Therapy intervention, which involves a 20-minute session of free-form Mandala coloring conducted one hour prior to their Objective Structured Clinical Examination (OSCE). The intervention is designed to reduce exam-related anxiety by promoting mindfulness, visual focus, and emotional self-regulation through creative expression.
  Interventions: Behavioral: Mandala Coloring
- Routine Academic Preparation (No Intervention): Participants in this group continue with their usual academic preparation and receive no additional interventions.

INTERVENTIONS:
Behavioral: Mandala Coloring — Participants in this group receive the Mandala Art Therapy intervention, a creative, mindfulness-based activity rooted in complementary and alternative medicine. The intervention is designed to reduce exam-related anxiety by fostering visual focus, emotional calm, and self-expression. The Mandala protocol includes the following components:
  * Distribution of printed Mandala outlines on A4 paper
  * Provision of six colored pencils (red, orange, yellow, green, blue, and purple)
  * A 20-minute individual coloring session in a quiet and relaxed setting
  * No prescribed patterns-participants color freely to encourage self-directed engagement The Mandala coloring session is conducted exactly one hour before the Objective Structured Clinical Examination (OSCE). The activity is supervised by the researcher to ensure a supportive and distraction-free environment. Participants are encouraged to concentrate on the process of coloring to promote psychological grounding and reduce pre-exam stress.
  Arms: Mandala Art Therapy

SUMMARY:
This randomized clinical trial aimed to evaluate the effectiveness of Mandala Art Therapy in reducing practical examination anxiety among undergraduate nursing students. The primary goal was to determine whether a brief Mandala coloring session prior to the Objective Structured Clinical Examination (OSCE) could significantly reduce students' state anxiety. The study focused on the therapeutic potential of this low-cost, non-invasive, and easily implemented intervention in academic settings.

The main research questions guiding the study were:

Does Mandala coloring reduce pre-examination anxiety among undergraduate nursing students?

Can Mandala Art Therapy be considered a feasible and effective complementary strategy for managing academic stress in clinical evaluation contexts?

To address these questions, participants were randomly assigned to either an experimental group, which engaged in a 20-minute Mandala coloring session before the OSCE, or a control group, which received no intervention beyond standard exam preparation. Pre- and post-intervention anxiety levels were measured using the Spielberger State-Trait Anxiety Inventory (STAI) to assess the impact of the intervention.

DETAILED DESCRIPTION:
Study Title:

The Influence of Mandala Art Therapy on Practical Examination Anxiety Among Undergraduate Nursing Students

Study Purpose:

The aim of this study was to evaluate the effectiveness of Mandala Art Therapy-a creative, mind-body intervention rooted in complementary and alternative medicine-in reducing practical examination (OSCE) anxiety among undergraduate nursing students. The intervention was implemented as part of a holistic approach to psychological well-being in a randomized, double-blind clinical trial.

Sample Size Determination:

The statistical population included undergraduate nursing students at Near East University. Out of 120 eligible students, 100 participants who met inclusion criteria were enrolled in the study after providing informed consent.

Participants were randomly assigned to either the experimental or control group using a simple randomization technique: 100 numbered cards were placed in a glass container and drawn alternately to assign participants to the two groups.

Based on parameters from a previous similar study (α = 0.05, power = 80%, S1 = 9.61, S2 = 10.4, μ1 = 42.03.5, μ2 = 47.7), the minimum required sample size was 48 per group. To allow for a 5% dropout rate, 50 students were ultimately placed in each group.

A double-blind design was used to reduce bias. The data collector was blinded to group allocations, and the statistician analyzing the data received anonymized variables coded as x1 and x2.

Tools of Data Collection:

A) Demographic Questionnaire:

Collected data on age, gender, marital status, and educational level.

B) Spielberger State-Trait Anxiety Inventory (STAI):

A validated 40-item tool assessing state and trait anxiety using a 4-point Likert scale. Higher scores indicated greater anxiety. The STAI has demonstrated strong psychometric properties, with a Cronbach's alpha of 0.96.

Intervention:

Experimental Group:Students participated in a 20-minute unstructured Mandala coloring session in a quiet room, one hour before the OSCE. Each student was provided with a Mandala outline and six colored pencils. The session aimed to foster mindfulness and reduce pre-exam anxiety.

Control Group:Students followed the standard university OSCE preparation routine without any additional intervention.

Implementation Phase:

The trial was conducted within the Nursing Department of Near East University. All students were briefed about the procedures and gave written informed consent. Mandala sessions were conducted in a distraction-free environment, and all participants completed STAI questionnaires before and after the intervention period.

Ethical Considerations: The study was approved by the Near East University Ethics Review Board (Approval No. NUE/2024/124-1854) and registered on ClinicalTrials.gov (NCT06571357). Ethical standards followed the Declaration of Helsinki (1964). All participants were informed of their right to withdraw at any time. Confidentiality and data protection were strictly maintained.

Statistical Analysis: All statistical analyses were conducted using SPSS version 25. The Kolmogorov-Smirnov test was used to assess normality. Data were analyzed using: Descriptive statistics (mean, SD, frequencies) Paired t-test (within-group pre-post comparison) Independent t-test (between-group comparison) Chi-square test (for categorical variables) A P-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. All students, both female and male, first semester of bachelor's degree, studying in nursing department of Near East University.
2. Not using other stress reduction methods including progressive muscle relaxation, drug therapy, etc. to control exam anxiety.
3. Those willing to participate in the project.

Exclusion Criteria:

1. Unwilling to continue cooperation in the project,
2. Using any psycho medicines (anti-depressants ...), mental health
3. Mourning, especially the death of loved ones or relatives in the 1st phase.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Practical Exam Anxiety Levels | Anxiety levels are measured at two time points-immediately before and immediately after the intervention session, conducted one hour prior to the OSCE
  The primary outcome measure assesses changes in anxiety levels related to the Objective Structured Clinical Examination (OSCE) among undergraduate nursing students. Anxiety is measured using the State-Trait Anxiety Inventory (STAI), a validated psychological instrument that evaluates both situational (state) and general (trait) anxiety. The STAI comprises two subscales with 20 items each, rated on a 4-point Likert scale. Higher total scores indicate greater levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Pouran Varvani Farahani, PhD, Principal Investigator — Department of Nursing, Faculty of Health Science, Cyprus International University
Locations (1):
- Near East University, Nicosia, KKTC (Turkish Republic of Northern Cyprus, Cyprus

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers